CLINICAL TRIAL: NCT00210275
Title: The Ontario Printed Educational Message (OPEM) Trial to Narrow the Evidence-practice Gap With Respect to Prescribing Practices of General and Family Physicians: a Cluster Randomized Controlled Trial
Brief Title: Ontario Printed Educational Materials (PEMs) for Physician Behaviour Change
Acronym: OPEMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Principal Investigator, Merrick Zwarenstein, Senior Scientist, Institute for Clinical Evaluative Sciences
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: MCT-67916
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Education, Medical, Continuing; Practice Patterns; Hypertension; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): Usual practice; no additional information provided.
- Printed Educational Message #1 (Experimental): Information about Angiotensin-converting enzyme inhibitors, hypertension treatment, and cholesterol lowering agents for diabetes
  Interventions: Behavioral: Printed Educational Message
- Printed Educational Message #2 (Experimental): Retinal screening for diabetes
  Interventions: Behavioral: Printed Educational Message
- Printed Educational Message #3 (Experimental): Diuretics for hypertension
  Interventions: Behavioral: Printed Educational Message

INTERVENTIONS:
Behavioral: Printed Educational Message — Three forms of printed educational materials (short or long educational messages and patient reminder notes)
  Arms: Printed Educational Message #1; Printed Educational Message #2; Printed Educational Message #3

SUMMARY:
The purpose of this study is to determine whether printed educational materials can change physician behaviour towards more evidence based decision-making.

DETAILED DESCRIPTION:
BACKGROUND:

There are gaps between what family practitioners do in clinical practice and the evidence-based ideal. The most commonly used strategy to narrow these gaps is the printed educational message (PEM); however, the attributes of successful printed educational messages and their overall effectiveness in changing physician practice are not clear. The current endeavor aims to determine whether such messages change prescribing quality in primary care practice, and whether these effects differ with the format of the message.

METHODS/DESIGN:

The design is a large, simple, factorial, unblinded cluster-randomized controlled trial. PEMs will be distributed with informed, a quarterly evidence-based synopsis of current clinical information produced by the Institute for Clinical Evaluative Sciences, Toronto, Canada, and will be sent to all eligible general and family practitioners in Ontario. There will be three replicates of the trial, with three different educational messages, each aimed at narrowing a specific evidence-practice gap as follows: 1) angiotensin-converting enzyme inhibitors, hypertension treatment, and cholesterol lowering agents for diabetes; 2) retinal screening for diabetes; and 3) diuretics for hypertension.For each of the three replicates there will be three intervention groups. The first group will receive informed with an attached postcard-sized, short, directive "outsert." The second intervention group will receive informed with a two-page explanatory "insert" on the same topic. The third intervention group will receive informed, with both the above-mentioned outsert and insert. The control group will receive informed only, without either an outsert or insert.Routinely collected physician billing, prescription, and hospital data found in Ontario's administrative databases will be used to monitor pre-defined prescribing changes relevant and specific to each replicate, following delivery of the educational messages. Multi-level modeling will be used to study patterns in physician-prescribing quality over four quarters, before and after each of the three interventions. Subgroup analyses will be performed to assess the association between the characteristics of the physician's place of practice and target behaviours.A further analysis of the immediate and delayed impacts of the PEMs will be performed using time-series analysis and interventional, auto-regressive, integrated moving average modeling.

ELIGIBILITY:
Inclusion Criteria:

* Family physicians or general practitioners in Ontario with >100 patients over 65 years of age in fee for service practice with >$50,000 billings to Ontario Health Insurance Plan (OHIP) in 2003

Exclusion Criteria:

* Physicians who have elected not to receive "informed". "informed" is a quarterly newsletter on evidence based practice produced by the Institute for Clinical Evaluative Sciences (ICES) and is the vehicle for delivery of the printed educational messages.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2005-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change in Behavioral intention related to referring patient for retinopathy screening | Two months and six months post intervention

SECONDARY OUTCOMES:
Change in Attitude (Theory of Planned Behaviour) | Two months and six months post intervention
Change in Subjective Norm (Theory of Planned Behaviour) | Two months and six months post intervention
Change in Perceived Behavourial Control (Theory of Planned Behaviour) | Two months and six months

CONTACTS AND LOCATIONS:
Overall Officials: Merrick F. Zwarenstein, MB, BCh, MSc, Principal Investigator — Institute for Clinical Evaluative Sciences